CLINICAL TRIAL: NCT00863122
Title: Exploration and Estimation of Intratumoral Concentration and Activity of Lapatinib in Vivo in Vestibular Schwannomas
Brief Title: Concentration and Activity of Lapatinib in Vestibular Schwannomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Children's Tumor Foundation (Other); GlaxoSmithKline (Industry); New York University (Other); Ohio State University (Other); House Research Institute (Other); Washington University School of Medicine (Other); Weill Medical College of Cornell University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: J0867; NA_00020841
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Vestibular Schwannoma; NF2; Neurofibromatosis 2; Acoustic Neuroma; Auditory Tumor
Keywords: Lapatinib; Tykerb; EGFR inhibitor; ErbB2 inhibitor; Pharmacokinetics
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2 | interventions — Lapatinib

ARMS (2):
- lapatinib (Experimental): Subjects will receive lapatinib for 10 days prior to surgery for vestibular schwannoma resection.
  Interventions: Drug: lapatinib
- control (No Intervention): Control subjects will not receive any intervention prior to surgery for vestibular schwannoma resection.

INTERVENTIONS:
Drug: lapatinib — 1500 mg lapatinib by mouth per day for 10 days
  Other Names: Tykerb
  Arms: lapatinib

SUMMARY:
Tumors can grow on the auditory nerves and can cause hearing loss. A common type of tumor that does this is a vestibular schwannoma (VS), or acoustic neuroma. These tumors are not cancerous. Most often, people have only one VS. Occasionally, people have more than one VS and may have a condition called neurofibromatosis type 2 (NF2).

Because VS can cause hearing loss, many people with VS will have treatment to preserve their hearing. This treatment usually involves surgery or radiation therapy. There are risks to these procedures, and sometimes they do not work to prevent hearing loss. Because surgery and radiation have risks and are not able to help everyone with VS, other methods of treatment are being explored. One area of exploration is looking to see if there is a drug that can be taken that might prevent the VS from growing larger and causing hearing loss, and might possibly even cause the VS to shrink in size.

This study is exploring whether a drug that is approved by the FDA and is currently used to treat breast cancer might also work to treat VS. This study will measure the amount of drug that travels from the bloodstream and arrives at the tumor. This drug is safe and has few side effects. If this drug is shown to reach the tumor, it might be used in the future to treat VS without needing surgery or radiation.

This study is recruiting people who are having surgery for VS. If you are going to have surgery to treat a VS, you may be eligible to participate.

DETAILED DESCRIPTION:
Neurofibromatosis type 2 (NF2) is a rare autosomal dominant genetic disorder with an incidence of approximately 1/40,000. The most common tumor type in NF2 is vestibular schwannoma and the majority of NF2 patients develop progressive hearing loss in adolescence or young adulthood due to bilateral vestibular schwannoma (VS). In addition to hearing loss, VS can cause significant morbidity, and in some cases mortality, due to brain stem compression.

Currently, the only accepted modality for treatment of VS in patients with NF2 is surgical resection. Although surgical resection is effective at tumor reduction, it is often associated with morbid complications such as hearing loss, facial palsy, CSF leaks, chronic headache and infection. In addition, the tumors often recur after surgery. Radiation therapy (RT) has been proposed as an alternative, however, its safety in the NF2 population has not been established and there is concern about long term efficacy. For a distinct population of NF2 patients, surgery and RT at not feasible and no additional therapy is currently available. Hence, a systemic therapy is needed.

Sporadic VS are common with roughly 3,000 new cases per year in the United States and a growing incidence in recent years. These tumors cause unilateral hearing loss, tinnitus, and vertigo. The primary treatment modality for these tumors is surgical resection or radiosurgery. Surgery is associated with the same complications listed above for NF2-related VS. Hence, RT is often offered in place of surgery. Although considered safe in sporadic VS, it may not have good long term efficacy and may complicate future procedures. Again, a systemic therapy that could control tumor progression obviating the need for an invasive procedure is needed.

As the understanding of tumor molecular biology continues to advance, there are an increasing number of attractive targets for VS growth inhibition. EGFR and ErbB2 have been identified as important targets for VS. In a study of 21 sporadic and 17 NF2-related VS samples, both EGFR and ErbB2 were found to be upregulated in the majority of tumors. In addition, an anti-ErbB2 monoclonal antibody reduced schwannoma cell proliferation in vitro. Collectively, this data suggests that abnormal signaling via EGFR and ErbB2 is a major contributor to tumor growth and progression in both sporadic and NF2-related VS, and that inhibition of this signaling pathway can result in decreased tumor growth. Although agents targeting these pathways are commercially available, there is little pre-clinical data to assist in prioritizing which agents to advance to clinical trials. Given the relative rarity of the disorder and the enormous patient, financial and time commitments an efficacy study requires, there is a need to carefully select agents for testing that have the best chance of success.

In this trial, we propose to assess the delivery of lapatinib, a commercially available inhibitor of ErbB2 and EGFR, to VS via tissue sampling at the time of clinically indicated surgery. Demonstrating that lapatinib reaches meaningful intratumoral concentrations is important data to recommend this drug above other small molecule inhibitors for efficacy trials for VS. The primary objective is to determine the steady state concentration of lapatinib in VS in patients with NF2 and in patients with sporadic VS. Patient who are planning to have surgical resection of their tumor for clinical indications will be given lapatinib for 15 days prior to resection. At the time of resection, VS tissue will be assessed for drug concentration and molecular markers of drug activity.

Demonstrating that lapatinib reaches meaningful concentrations within VS would support selecting this agent for investigation in efficacy studies for VS, and tissue-based molecular studies will provide corollary information about the behavior of VS in general and about lapatinib specifically in VS tissue. This may further our understanding of the pathophysiology of VS, the similarities and differences between NF2-related and sporadic VS, and inform the design of subsequent efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for NF2 including presence of bilateral VS or idiopathic VS without evidence of genetic syndrome.
* VS surgery determined clinically necessary by the treating physician and scheduled within 4 weeks.
* Normal cardiac left ventricular ejection fraction (LVEF) by multiple-gated acquisition (MUGA) scan or transthoracic echocardiogram.
* Karnofsky performance status 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Must have the following hematologic, renal and liver function: Absolute neutrophil count ≥ 1,000/mm³ (unsupported); platelet count ≥ 75,000/mm³ (unsupported); hemoglobin ≥ 8 g/dL (transfusion support allowed); Creatinine ≤ 1.5 times upper limit of normal (ULN) OR glomerular filtration rate ≥ 70 ml/min; Bilirubin ≤ 1.5 times ULN; ALT ≤ 2.5 times ULN.
* Be able to provide written informed consent.
* Any neurologic deficits must be stable for ≥ 1 week.
* Be able to swallow tablets.
* Subjects with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test.
* Suspend the use of P450 inducing or P450 suppressing agents for a minimum of 10 days prior to starting lapatinib.

Exclusion Criteria:

* Serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Pregnant or breast-feeding.
* Receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents, radiation or immunotherapy) within 4 weeks of the first dose of the study drug.
* Concurrent or prior malignancy, other than curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Subjects who have been free of disease (any prior malignancy) for five years are eligible for this study.
* Received cytochrome P450-inducing anticonvulsants (EIADs; e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) or similar agents (e.g., rifampin) or P450 inhibiting agents (Ketoconazole, Itraconazole, Clarithromycin, Atazanavir, Indinavir, Nefazodone, Nelfinavir, Ritonavir, Saquinavir, Telithromycin, Voriconazole) within 10 days prior to starting lapatinib.
* Significant gastrointestinal disorder(s)(e.g., Crohn's disease, ulcerative colitis, extensive gastric resection).
* Neurologic deficits that are rapidly progressing.
* Known cardiac disease (either arrhythmia or congestive heart failure) requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaishri O Blakeley, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - House Reserach Institute, Los Angeles, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Weil Cornell Medical College, New York Presbyterian Hospital, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients undergoing surgery for vestibular schwannoma resection who met eligibility criteria were invited to participate
Pre-assignment Details: Patients could enroll on control (no drug) or lapatinib arms. 20 people were consented for the the lapatinib arm, but one patient withdrew consent prior to completion of eligibility screening and enrollment. So 19 patients enrolled on the lapatinib arm.
Groups:
- Lapatinib: Subjects received lapatinib 1500 mg by mouth for 10 days prior to surgery for vestibular schwannoma resection.
- Control: Control subjects did not receive any intervention prior to surgery for vestibular schwannoma resection.
Period: Overall Study
Arm/Group | Lapatinib | Control
Started | 19 | 7
Completed | 19 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lapatinib: Subjects received lapatinib for 1500 mg by mouth daily for 10 days prior to surgery for vestibular schwannoma resection
- Total: Total of all reporting groups
Arm/Group | Lapatinib | Control | Total
Number analyzed (Participants) | 19 | 7 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 7 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 44 [20 to 60] | 40 [30 to 61] | 43.5 [20 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 19 | 7 | 26
Karnofsky Performance Status (KPS) [Median (Full Range); unit: units on a scale (percent)] — KPS is a physician-reported outcome measuring an individual's functional impairment. Scores range from 0% (death) to 100% (normal no complaints; no evidence of disease).
  Specific to these results, 70% represents an ability to care for self; unable to carry on normal activity or to do active work, and 90% represents an ability to carry on normal activity; minor signs or symptoms of disease. Population: Per protocol, KPS was not recorded for control participants. Control participants agreed to donate tissue only. No clinical data was collected.
  units on a scale (percent)
    number analyzed (Participants) | 19 | 0 | 19
    (all) | 90 [70 to 100] |  | 90 [70 to 100]
Patients with a diagnosis of NF2 [Number; unit: participants] | 9 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Median Steady-state Lapatinib Plasma Concentrations at the Time of Surgical Resection
Description: Steady-state plasma concentrations of lapatinib (ng/mL) at time of surgery, 10-13 days from starting drug.
Time Frame: At time of surgery, 10-13 days from starting drug.
Population: In the lapatinib group, 10 tissue and plasma samples were lost from analysis due to a freezer failure during a natural disaster denaturing the samples. 1 blood sample was contaminated, but tissue was available. Control group did not get any drug. A total of 8 participants of 19 given drug had data for analysis.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Lapatinib
Number analyzed (Participants) | 8
ng/mL | 3149 [786 to 5830]

2. Primary Outcome: To Assess Whether Lapatinib Can Reach a Minimum Tumor Concentration Level of >3uM in VS After Oral Dosing.
Description: Count of tissue samples with lapatinib concentration >3uM
Time Frame: one year
Population: In the lapatinib group, 10 tissue and plasma samples were lost from analysis due to a freezer failure during a natural disaster denaturing the samples. Nine samples were available for tissue concentration assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 9
Participants | 7

3. Secondary Outcome: Assess the Level of ErbB2 Phosphorylation in VS.
Description: Assessed number of samples with high expression of phospho-ErbB2 in tissue at time of surgery
Time Frame: at time of surgery
Population: 10 lapatinib participants and 3 control participants did not have adequate tissue for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control subjects will not receive any intervention prior to surgery for vestibular schwannoma resection. Control subjects donate tissue at the time of surgery.
Arm/Group | Lapatinib | Control
Number analyzed (Participants) | 9 | 4
Participants | 5 | 2

4. Secondary Outcome: Assess Markers of Tumor Proliferation and Cell Death in VS After Exposure to Lapatinib.
Time Frame: At time of surgery
Population: The experiment to assess this outcome measure failed and no interpretable data could be collected.
Arm/Group | Lapatinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Explore the Difference in the Concentration of Lapatinib Achieved in NF2-related Versus Idiopathic VS.
Description: A comparison in the median lapatinib concentration (ng/g) in vestibular schwannomas associated with neurofibromatosis type 2 and sporadic vestibular schwannomas
Time Frame: one year
Population: Of the nine participants in the lapatinib who had tumor available for analysis, four had a vestibular schwnannoma associated with a diagnosis of neurofibromatosis type 2 (NF2); five had sporadic vestibular schwannomas.
Measure: Median (Full Range); unit: ng/g
Groups:
- NF2 Associated VS: Participants with vestibular schwannomas associated with a diagnosis of neurofibromatosis type 2
- Sporadic VS: Participants with sporadic vestibular schwannomas (i.e. not associated with a diagnosis of neurofibromatosis type 2)
Arm/Group | NF2 Associated VS | Sporadic VS
Number analyzed (Participants) | 4 | 5
ng/g | 8367 [314 to 17821] | 4502 [1737 to 11712]

6. Secondary Outcome: Perform NF2 Gene Mutation Analysis Via Exon Scanning and MLPA as Well as Protein Expression in All VS and Explore Differences Between Sporadic and NF2 Related VS.
Description: Due to the sample sizes, a comparison between sporadic and NF2-related vestibular schwannomas could not be made. Instead we report the mutational status.
Time Frame: at time of surgery
Population: 6 of the 7 participants had sporadic VS; 1 of 7 had NF2-associated VS. As such, we were unable to explore differences between the groups.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Tissue Available for Gene Mutation Analysis: Seven participants had successful NF2 gene mutation analysis via exon scanning and MLPA.
Arm/Group | Participants With Tissue Available for Gene Mutation Analysis
Number analyzed (Participants) | 7
Participants
  Hemizygous deletion in NF2 gene | 4
  Homozygous deletion in NF2 gene | 1
  No deletion in NF2 gene | 2

ADVERSE EVENTS:
Description: Zero participants were At Risk from the Control arm since they did not receive any intervention.
Groups:
- Control: Control subjects will not receive any intervention prior to surgery for vestibular schwannoma resection. Control subjects donate tissue at the time of surgery. AEs were not collected in this group as there was no study intervention (i.e. they did not take the drug).
Arm/Group | Lapatinib | Control
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 12/19 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib (N=19) | Control (N=0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
A total of 10 tissue and 11 plasma samples donated by participants receiving lapatinib and 2 tissue samples from control participants were lost from analysis due to freezer failure denaturing the samples. This substantially reduced the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less